CLINICAL TRIAL: NCT03143517
Title: CALFE Stool Sample Collection Protocol
Brief Title: Fecal Calprotectin Collection Protocol
Acronym: CALFE
Status: Completed | Type: Observational
Sponsor: DiaSorin Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CALFE Sample Collection C-001
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Ulcerative Colitis; Crohn Disease; Indeterminate Colitis; Chronic Diarrhea; Celiac Disease; Diverticulitis; Abdominal Pain; Distension; Weight Loss; Food Intolerance; Constipation
Keywords: Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Ulcerative Colitis; Crohn Disease; Indeterminate Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Colitis, Ulcerative; Crohn Disease; Celiac Disease; Diverticulitis; Abdominal Pain; Dilatation, Pathologic; Weight Loss; Food Intolerance; Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Stool
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Inflammatory Bowel Disease (IBD): A stool sample will be collected from adult subjects with Inflammatory Bowel Disease (IBD), confirmed by endoscopy and histologic examination.
  Interventions: Diagnostic Test: Stool collection
- Irritable Bowel Syndrome (IBS): A stool sample will be collected from adult subjects with adult subjects with Irritable Bowel Syndrome meeting the Rome III criteria.
  Interventions: Diagnostic Test: Stool collection
- Other GastroIntestinal (GI) Disorders: A stool sample will be collected from adult subjects with adult subjects with gastrointestinal disorders other than IBD or IBS.
  Interventions: Diagnostic Test: Stool collection

INTERVENTIONS:
Diagnostic Test: Stool collection — Stool sample collected by a subject who have been diagnosed with IBD, IBS or other GI disorder. The stool sample is tested in a laboratory where fecal calprotectin levels are quantified.

SUMMARY:
The primary objective is to obtain stool samples from subjects diagnosed with , and displaying signs and/or symptoms of IBD and/or IBS will be evaluated in this study. Eligible subjects require a diagnostic colonoscopy with possible biopsy and clinical evaluation.

DETAILED DESCRIPTION:
Stools will be collected and tested, at a later date, in a clinical performance study with an investigational Calprotectin assay. This study will be coordinated by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of either gender and ≥ 4 years of age.
* Subject is showing signs and symptoms of IBD and/or IBS.
* Diagnosis of IBD, IBS or other gastrointestinal disorder is performed by colonoscopy.
* Subject or authorized legal representative is willing and able to sign the IRB approved Informed Consent form or able to provide Informed Consent in accordance with 21 CFR 50 CFR 50 Subpart B.
* Subject is able to understand and follow study sample collection procedure.

Exclusion Criteria:

* Subject has undergone a surgical resection or diversion procedure.
* Subject is currently taking NSAIDS (non-steroidal anti-inflammatory drugs, i.e. ibuprofen, Advil, Motrin, Naproxen, Aleve including regular dose and low dose aspirin) within 7 days of colonoscopy and sample collection.
* Subject who has taken immunomodulators or biologic therapies within the previous 6 months of colonoscopy and sample collection.
* Subject who is currently pregnant or lactating.
* Subject is unable or unwilling to follow informed consent.
* Inability or unwilling to perform required study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects and belonging to the target population, i.e. patients diagnosed with IBD, specifically CD, UC, or IC, patients diagnosed with IBS, and patients diagnosed with other gastrointestinal diseases, e.g. Celiac Disease, Diverticular Disease, Chronic Diarrhea and Recurrent Abdominal Pain (RAP).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Calprotectin Stool Collection | Through Study Completion, an average of 1 year
  In vitro diagnostic (IVD) device performance

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - One (1) Location in Dothan, Alabama, Dothan, Alabama
  - One (1) Facility in Arkansas, Little Rock, Arkansas
  - One (1) Location in California, Mission Hills, California
  - One (1) Location in Colorado Springs, Colorado, Colorado Springs, Colorado
  - One (1) Location in Lauderdale Lakes, FL, Lauderdale Lakes, Florida
  - One (1) Location in Maitland, FL, Maitland, Florida
  - One (1) Location in Miami, Florida, Miami, Florida
  - One (1) Location in St. Augustine, FL, Saint Augustine, Florida
  - One (1) Location in Atlanta, GA, Atlanta, Georgia
  - One (1) Location in Minneapolis, MN, Minneapolis, Minnesota
  - One (1) Location in New York, New York, New York, New York
  - One (1) Location in North Carolina, Asheville, North Carolina
  - One (1) Location in Greenville, SC, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided